CLINICAL TRIAL: NCT00778999
Title: A Randomized, Open-Label Clinical Trial to Identify Predictive Factors for Controlled Ovarian Stimulation Using a Fixed Daily Dose of 200 IU Recombinant FSH in GnRH Antagonist Regimen With or Without Oral Contraceptive Scheduling
Brief Title: Predictive Factors for Ovarian Stimulation Using a Fixed Daily Dose of 200 IU Recombinant FSH (Study 142003)(P05696)
Acronym: Xpect
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05696; 142003; NCT00628641 (obsolete NCT alias)
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Results first posted 2009-08-12 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Desogestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Contraceptive (Active Comparator): Use of oral contraceptive pills prior to controlled ovarian stimulation
  Interventions: Drug: Marvelon
- Non-Oral Contraceptive (No Intervention): No use of oral contraceptive pills prior to controlled ovarian stimulation

INTERVENTIONS:
Drug: Marvelon — oral contraceptive 1 tablet daily for 14 to 21 days
  Arms: Oral Contraceptive

SUMMARY:
The success of assisted reproductive technologies (ART) is critically dependent on optimizing protocols for controlled ovarian stimulation to provide adequate numbers of good quality oocytes and embryos. This optimization is mainly valuable to a group of infertility patients (9%-24%) who respond poorly to Controlled Ovarian Stimulation(COS). It is also important for an additional 2.6% of the infertility patients who manifest a high response to gonadotropin and are at risk for hyperstimulation syndrome, a life-threatening situation. Extensive research was carried out and led to the introduction of GnRH antagonist, as an alternative to Gonadotropin Releasing Hormone (GnRH) agonist, for the prevention of premature Luteinizing Hormone (LH) surges. Further research to optimize the GnRH antagonist regimen concluded that a daily treatment with 200 IU of recombinant Follicle Stimulating Hormone (recFSH) in a GnRH antagonist regimen is safe, well tolerated and results in a good clinical outcome. This protocol is now frequently applied in the US and Europe.

Predicting a woman's response (based on the assessment of ovarian reserve) to COS is useful in determining individualized clinical management strategies for low and high responders and thus avoiding cancellation. Such prediction when based on reliable scientific evidence is valuable in consulting patients about their chances of success. A large number of studies have been performed, which used certain clinical, ultrasonographic and hormonal markers (called predictive factors), to try to optimize a COS protocol for patients who were down-regulated with a long GnRH agonist protocol. Prospective trials of predictive models have also been used to adjust the starting dose of FSH to prevent a too low or too high ovarian response. To date, however, none have been performed for women undergoing ovarian stimulation with a GnRH antagonist protocol.

The primary objective of this randomized, open-label, multicenter clinical trial was to identify one or more factors capable of predicting ovarian response in women treated with a daily dose of 200 IU recFSH in a GnRH antagonist protocol. Since many ART centers now use oral contraceptives as a means to schedule patients stimulated with recFSH and a GnRH antagonist for assisted reproduction, the trial evaluated also whether intervention with oral contraceptives affects the accuracy of predictive models for ovarian response.

ELIGIBILITY:
Inclusion Criteria:

* Females of couples with an indication for In Vitro Fertilization (IVF) and/or Intracytoplasmic Sperm Injection (ICSI) scheduled for their first COS treatment cycle
* Females >18 and <=39 years of age at the time of signing informed consent
* Body Mass Index (BMI) <= 32 kg/m^2
* Normal menstrual cycle length; 24-35 days
* Availability of ejaculatory sperm (use of donated and/or cryopreserved sperm is allowed)
* Willing and able to sign informed consent

Exclusion Criteria:

* History of/or any current endocrine abnormality
* Less than 2 ovaries or any other ovarian abnormality (inc.>10mm endometrioma)
* Presence of unilateral or bilateral hydrosalpinx
* Presence of any clinically relevant pathology affecting the uterine cavity or fibroids >= 5cm
* History of recurrent miscarriage (3 or more, even when unexplained)
* FSH or LH > 12 IU/L as measured by a local laboratory (sample taken during the early follicular phase: menstrual day 2-5)
* Any clinically relevant abnormal laboratory value (FSH, LH, estradiol (E2), Progesterone (P), total Testosterone (T), prolactin, Thyroid Stimulating Hormone (TSH), blood biochemistry, hematology and urinalysis) based on a sample during the screening phase.
* Contraindications for the use of gonadotropins (tumors, pregnancy, lactation, undiagnosed vaginal bleeding, hypersensitivity, ovarian cysts)
* Contraindications for the use of oral contraceptive pills (history of (h/o) thromboembolism, breast cancer, undiagnosed vaginal bleeding)
* Recent history of/or current epilepsy, Human Immunodeficiency Virus (HIV) infection, diabetes, cardiovascular, gastrointestinal, hepatic, renal or pulmonary disease
* Abnormal karyotyping of the patient or her partner (if karyotyping is performed)
* History or presence of alcohol or drug abuse within 12 months of signing the consent
* Use of hormonal preparations within one month prior to randomization
* Hypersensitivity to any of the concomitant medication prescribed as part of the treatment regimen in this protocol
* Administration of investigational drugs within three months prior to signing the informed consent

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 442 (Actual)
Dates: Start 2006-10-01 (Actual); Primary Completion 2008-07-24 (Actual); Study Completion 2008-07-24 (Actual)

REFERENCES:
- [Derived] Broekmans FJ, Verweij PJ, Eijkemans MJ, Mannaerts BM, Witjes H. Prognostic models for high and low ovarian responses in controlled ovarian stimulation using a GnRH antagonist protocol. Hum Reprod. 2014 Aug;29(8):1688-97. doi: 10.1093/humrep/deu090. Epub 2014 Jun 5. PMID 24903202
- [Derived] Andersen AN, Witjes H, Gordon K, Mannaerts B; Xpect investigators. Predictive factors of ovarian response and clinical outcome after IVF/ICSI following a rFSH/GnRH antagonist protocol with or without oral contraceptive pre-treatment. Hum Reprod. 2011 Dec;26(12):3413-23. doi: 10.1093/humrep/der318. Epub 2011 Sep 27. PMID 21954280

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Contraceptive | Non-Oral Contraceptive
Started | 223 | 219
Completed | 195 | 185
Not Completed | 28 | 34
Not completed — Discontinuation: no embryo transfer | 14 | 14
Not completed — Did not receive recFSH | 14 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Contraceptive | Non-Oral Contraceptive | Total
Number analyzed (Participants) | 223 | 219 | 442
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 223 | 219 | 442
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 223 | 219 | 442
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Oocytes
Description: The total number of oocytes on the Day of oocyte pick-up is an indication of ovarian response
Time Frame: 12 weeks
Population: Intent-to-treat, defined as all randomized subjects who received recombinant follicle stimulating hormone
Measure: Mean (Standard Deviation); unit: Number of oocytes
Arm/Group | Oral Contraceptive | Non-Oral Contraceptive
Number analyzed (Participants) | 209 | 199
Number of oocytes | 12.4 (6.7) | 12.1 (7.7)

2. Secondary Outcome: Number of Mature Oocytes
Description: This is not a prespecified key secondary outcome; therefore, results will not be disclosed.
Time Frame: 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Number of Follicles on Stimulation Day 8
Description: This is not a prespecified key secondary outcome; therefore, results will not be disclosed.
Time Frame: 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Number of Follicles on Day of hCG
Description: This is not a prespecified key secondary outcome; therefore, results will not be disclosed.
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Number of Fertilized (2PN) Oocytes
Description: This is not a prespecified key secondary outcome; therefore, results will not be disclosed.
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Number of Good Quality Embryos
Description: This is not a prespecified key secondary outcome; therefore, results will not be disclosed.
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Oral Contraceptive | Non-Oral Contraceptive
Serious Adverse Events (participants affected / at risk) | 10/209 | 9/199
Other Adverse Events (participants affected / at risk) | 88/209 | 81/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Contraceptive (N=209) | Non-Oral Contraceptive (N=199)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Antepartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2)
Retroplacental haematoma (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 2 (2) | 3 (3)
Abortion induced (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Contraceptive (N=209) | Non-Oral Contraceptive (N=199)
Nausea (Gastrointestinal disorders) | 8 (8) | 15 (18)
Procedural pain (Injury, poisoning and procedural complications) | 53 (55) | 45 (45)
Headache (Nervous system disorders) | 17 (23) | 12 (12)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 12 (12)
Antepartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 11 (14) | 9 (13)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 5 (5) | 11 (11)
Pelvic discomfort (Reproductive system and breast disorders) | 20 (21) | 14 (16)
Pelvic pain (Reproductive system and breast disorders) | 18 (20) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor recognizes the right of the investigator(s) to publish, but all communication concerning the clinical trial must be based on data validated and released and will first be submitted to the Sponsor for written consent, which shall not be withheld unreasonably. Sponsor is free to use the data for publication. The investigator(s) may be invited to be co-author(s). In any communication concerning this clinical trial, the author(s) of this protocol will be included in the list of authors.